CLINICAL TRIAL: NCT05342961
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial to Evaluate the Safety and Efficacy of Spinous Balloon Dilatation Catheter (Plastic-BladeTM) in the Treatment of Coronary Artery Disease
Brief Title: Safety and Efficacy of Spinous Balloon Dilatation Catheter in CAD Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CCRF Inc., Beijing, China (Industry)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KDL-SUF-2021001
Record Dates: First submitted 2022-03-15; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Masking Description: During the study, it is difficult for researchers, operators and patients to blind the method due to objective reasons.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinous balloon dilatation catheter(Plastic-Blade) (Experimental): Patients with CAD will be treated with spinous balloon dilatation catheter(Plastic-Blade).
  Interventions: Procedure: spinous balloon dilatation catheter (Plastic-Blade)
- spinous balloon dilatation catheter(lacrosse NSE) (Experimental): Patients with CAD will be treated with spinous balloon dilatation catheter(lacrosse NSE)
  Interventions: Procedure: spinous balloon dilatation catheter(lacrosse NSE)

INTERVENTIONS:
Procedure: spinous balloon dilatation catheter (Plastic-Blade) — To treat Coronary artery disease
  Arms: spinous balloon dilatation catheter(Plastic-Blade)
Procedure: spinous balloon dilatation catheter(lacrosse NSE) — To treat Coronary artery disease
  Arms: spinous balloon dilatation catheter(lacrosse NSE)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of spinous process balloon dilation catheter (Plastic-Blade) in coronary vascular diseases, which is not inferior to the similar product on the market - coronary spinous process balloon dilation catheter (lacrosse NSE) produced by Goodman Co., Ltd..

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, controlled and non inferiority designed clinical trial. A total of 160 subjects with CAD from 8 centers will be randomized 1:1 to each group. All subjects evaluated the immediate lumen acquisition immediately after operation and the MACE of 30 ± 7 days after operation. The primary endpoint is the acquisition of lumen immediately after operation. The effectiveness of balloon was evaluated. The safety of balloon was evaluated by adverse events during operation.Clinical follow-up will be conducted at operation, discharge and 30 ± 7 days after operation. The target lesions included the following : opening lesions, bifurcation lesions, calcification lesions and fibrosis lesions; Diameter stenosis ≥ 70% (visual) with evidence of ischemia; Localized lesions with TIMI ≥ 1; RVD=2.00 and 4.00mm , and the vascular segment is suitable for balloon dilatation in anatomical structure。

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-75 years
* 2.Stable or unstable angina, or previous myocardial infarction, or Asymptomatic ischemia judged by clinician ,Target vascular diameter: 2.00-4.00mm ,Coronary artery stenosis stenosis ≥ 70% by visual inspection, or ≥ 50% with evidence of ischemia, TIMI blood flow≥ 1,the operator judge that the patient needs spinous balloon to treat.
* 3. Paticipant can understand the study ,voluntarily participate in and sign the informed consent form,and accept scheduled follow-up.

Exclusion Criteria:

Patient related:

* 1.Pregnant and breast-feeding women or intention to be pregnant.
* 2.Subjects with MI within one week, or more than one week after the onset of MI,but TNI or TNT have not returned to normal.
* 3.The spinous balloon failed to pass through the stenosis after small balloon dilation , and the lesion need to be rotary grinded.
* 4. Non-target vessel did not be dealed with successful before dealing with target vessel, or non-target vascular lesion number is more than three.
* 5.Serious heart failure（NYHA IV）
* 6.Severe renal failure（Cr>443uMol/L) or patients undergoing hemodialysis.
* 7.Patient with heart transplant.
* 8.Patient with CABG.
* 9.Patients with hemodynamic instability or shock symptoms.
* 10.Life expectancy less than one year.
* 11.Expected to undergo surgery within one month.
* 12.Patients with bleeding tendency, history of active gastrointestinal ulcer, contraindications of antiplatelet or anticoagulant treatment, cannot receive anticoagulant treatment, and patients have hemorrhagic stroke within six months.
* 13.Allergy to heparin and contrast agent.
* 14.The illness of the patient make the treatment and evaluation difficult.
* 15.Those who have participated in other drug or medical device trials have not reached main research endpoint.
* 16.Clinicians estimated that the risk of intervention is very high or the patient should be excluded for other reasons.
* 17.Poor of compliance

Lesion related:

* 18.Lesions of LAD or with a distance of ≤ 2mm beyond LAD.
* 19.Angiogram showed thrombus.
* 20.CTO,and TIMI blood flow=0,
* 21.Coronary artery spasm
* 22.Lesions of LAD without bypass surgery or collateral circulation protection.
* 23.The doctor considered the patient unfit for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-05-16 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Immediate lumen acquisition | during the procedure
  The difference of the minimum diameter of the target lesion before and after balloon dilatation in the test or control group measured by QCA.

SECONDARY OUTCOMES:
Rate of device success | during the procedure
  Proportion of patients who meet the success criteria. Success criteria be defined as the residual stenosis of the target lesion is less than 50% after balloon dilatation and the balloon delivery system is successfully withdrawn
Rate of clinical success | from procedure to discharge ( to the 7th day after procedure)
  Based on device success, no patient occurred composite endpoint (PoCE) during hospitalization
Incidence of related complications | 30 days after balloon dilatation
  Including acute occlusion, vasospasm, vascular rupture, branch or collateral occlusion, subacute stent thrombosis, intimal tear, dissection, etc.
% change of clinically meaningful laboratory tests | 30 days after procedure
  Record the change of clinically meaningful laboratory tests
Number of adverse events | 30 days
  Adverse events occurred during balloon dilatation, after balloon dilatation to 30 ± 7 days after discharge
Number of device related composite endpoint | 30 days
  Including TLF, Cardiac Death, TV-MI and ID-TLR
Number of patient oriented composite endpoint | 30 days
  Including all cause death, MI, TLR, TVR, Revascularization of any coronary arteries and thrombus at the lesion.
Total time of device operation performance | 30 days
  Push capacity, passing capacity and withdrawal capacity

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, MD.,Ph D., Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital

IPD SHARING:
Plan to Share IPD: No